CLINICAL TRIAL: NCT00277654
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Risperidone Monotherapy in Ambulatory Bipolar Disorder With Concurrent Moderately Severe Anxiety and Lifetime Panic or Generalized Anxiety Disorder
Brief Title: Study of Risperidone Monotherapy in Ambulatory Bipolar Disorder With Concurrent Moderately Severe Anxiety and Lifetime Panic or Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Janssen Pharmaceuticals (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RIS-PAD-402
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Bipolar Disorder; Anxiety Disorder
Keywords: Bipolar Disorder with Concurrent Moderately Severe Anxiety and Lifetime Panic or Generalized Anxiety Disorder
MeSH Terms: conditions — Bipolar Disorder; Anxiety Disorders; Generalized Anxiety Disorder | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Risperidone (Active Comparator)
  Interventions: Drug: Risperidone
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — risperidone 0.5mg up to 4mg daily vs. placebo
  Other Names: Risperidal

SUMMARY:
The purpose of this research study is to evaluate the safety, tolerability, and efficacy (how well the drug works) of risperidone compared to placebo (an inactive drug) in the treatment of bipolar disorder with panic disorder or generalized anxiety disorder. Risperidone is currently approved by the United States Food and Drug Administration (FDA) for the treatment of schizophrenia and bipolar mania. Risperidone is not currently FDA approved for the treatment of bipolar hypomania with or without panic disorder or generalized anxiety disorder (the condition being investigated in this study).

DETAILED DESCRIPTION:
Methods and Procedures:

This is a randomized, double-blind, placebo controlled, parallel-group, 3 site, 8-week trial of risperidone monotherapy in outpatient subjects with a lifetime bipolar I, II, or not otherwise specified (NOS) disorder, a lifetime panic or generalized anxiety disorder, and current, at least moderately, severe anxiety symptoms. Approximately 90 subjects will be enrolled to obtain 60 subjects who complete the 8-week trial. Subjects will be randomized to risperidone or placebo in a 1:1 ratio. No concomitant psychotropic medication will be allowed except for as needed (prn) lorazepam during the first two weeks for the management of affective and anxiety symptoms, and prn zolpidem and zaleplon throughout the study for the management of insomnia. Throughout the study, psychiatric scales will be used to assess psychiatric symptoms and the presence of treatment-emergent adverse events will be monitored and recorded.

Medication Dosing:

Risperidone will be administered at an initial dose of 0.5 to 1 mg/day and will be titrated upward to a dose considered optimal by the investigator based on the subject's clinical response and adverse events, but not to exceed 2.0 mg/day by the end of the second week. Subsequently, risperidone may be increased based on clinical response and tolerability to a maximum of 4.0 mg/day. As needed study-prescribed (prn) use of lorazepam will be allowed for the management of affective and anxiety symptoms for the first two weeks of the study; a maximum of 2 mg per day will be allowed during the first week, and a maximum of 1 mg per day will be allowed during the second week. During the second week, the subject must be tapered off the lorazepam. For the final six weeks of the study, no lorazepam will be permitted. Zolpidem (10-20 mg/day) or zaleplon (10-20 mg/day) will be allowed for management of insomnia, and benztropine (0.5 - 3.0 mg/day) will be allowed for management of extrapyramidal symptoms. The latter three agents will be permitted throughout the study.

From week 2 on, any medications with psychotropic effects are prohibited.

Screening Visit(s):

The Screening Period will last a minimum of 2 to a maximum of 30 days. At the first screening visit (Visit 0), informed consent will be obtained. The Mini International Neuropsychiatric Interview (MINI), with the Manic Module from the MINI plus, will be performed to establish whether the patient meets DSM-IV criteria for bipolar disorder I, II, or NOS, and for panic disorder or generalized anxiety disorder. For generalized anxiety disorder, the portion of Criterion F - that stipulates "the disturbance does not occur exclusively during a mood disorder" will be suspended. The CGI-BP and the CGI-S will be performed to establish the severity of bipolar affective symptoms and anxiety symptoms, respectively. Subjects will keep a mood chart in between visits to help them follow their affective and anxiety symptoms. The subject's bipolar symptoms must be evaluated as no more than moderately severe (defined as a CGI-BP < 4), and his/her anxiety symptoms must be evaluated as at least moderately severe (a CGI-S of > 4) for him/her to be able to continue in the screening process and enter the randomized phase. Medical history will be reviewed, a physical exam performed, electrocardiogram (EKG) and laboratory studies (complete metabolic profile, CBC with differential and platelets, urinalysis, pregnancy test, and urine drug screen) will be obtained. Based on these evaluations, it will be determined whether subjects meet entry criteria; subjects meeting these criteria will continue in the screening process.

Baseline Visit (last Screening Visit):

At baseline (Visit 1), subjects whose screening evaluations continue to meet all inclusion/exclusion criteria may enter the study and be randomized. These evaluations will include repeating the Clinical Global Impression modified for bipolar illness (CGI-BP) and the Clinical Global Improvement Scale for anxiety symptoms (CGI-S) to ensure the subject continues to have no more than moderately severe bipolar affective symptoms and at least moderately severe anxiety symptoms. Baseline ratings will include: the Sheehan Panic Anxiety Scale-Clinician Rated (SPAS-C); the Hamilton Anxiety Scale (HAM-A) to assess anxiety symptoms; the Young Mania Rating Scale (YMRS) to assess manic symptoms; and the Inventory for Depressive Symptoms (IDS) (long form) to assess depressive symptoms. Subjects will also be evaluated with the CGI-BP, and the Sheehan Disability Scale (SDS). The Panic-Agoraphobic Spectrum-Self-Report (PAS-SR) will be used to assess the lifetime presence of core and related features of panic disorder. (Subjects who score > 35 on the PAS-SR will be classified a-priori as having panic spectrum symptoms [PSS]). The Family Impact Scale (FIS) will be administered. The Abnormal Involuntary Movement Scale (AIMS), Simpson Angus Scale (SAS), and Barnes Akathisia Rating Scale (BARS) will be administered to assess for extrapyramidal symptoms. Blood pressure, pulse, height, and weight, will be measured. Study medication will be dispensed by the Physician Investigator in the form of 0.5 mg capsules. The dose range of risperidone will be 0.5 to 4 mg/day.

Treatment Period:

Study visits will occur every week through the eight weeks of treatment. It is expected that risperidone will be gradually increased to an optimal dose during the first month of treatment. The following procedures will be completed at each visit.

1. Collect unused risperidone, perform study drug accountability, and record dosage of study drug used. A subject's unused study medication can be re-dispensed back to the subject.
2. Review mood chart and administer Clinician Global Improvement on anxiety symptoms -21 point scale (CGI-I-21), Patient Global Improvement on anxiety symptoms -21 point scale (PGI-21), SPAS-C, HAM-A, YMRS, IDS, CGI-BP, and SDS ratings.
3. Assess and record adverse events.
4. Perform AIMS, SAS, and BARS.
5. Obtain blood pressure, pulse, and weight.
6. Record concomitant medication use (from mood chart)
7. Adjust risperidone dose (if necessary) and dispense study drug.

Final Evaluation (week 8) or Early Termination:

The following evaluations will be conducted at the completion of, or early withdrawal from, the 8-week treatment phase. All psychiatric evaluations and all other final study procedures (including a repeat physical exam, EKG, and laboratory studies) will be completed prior to the discontinuation of risperidone. The evaluations to be performed are:

* Collect unused risperidone, perform study drug accountability, and record dosage of study drug used.
* Review mood chart and perform CGI-21, SPAS-C, HAM-A, YMRS, IDS, CGI-BP, PGI-21, and SDS ratings.
* Repeat PAS-SR
* Repeat FIS
* Assess and record adverse events.
* Obtain blood pressure, pulse, weight, and determine BMI.
* Perform physical examination, AIMS, SAS, BARS.
* Obtain laboratories (complete metabolic profile, CBC with/differential and platelets, urinalysis, pregnancy test, and urine drug screen).
* Repeat EKG.
* Record concomitant medication use (from mood chart)
* Adjust risperidone dose (if necessary) and prescribe drug (if subject has responded and chooses to continue on risperidone), or dispense risperidone taper for discontinuation (if subject has not responded or if subject chooses to discontinue risperidone for any reason).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older.
2. Subjects must have lifetime bipolar I, II, or NOS disorder as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria.
3. Subjects must have lifetime panic disorder or generalized anxiety disorder (GAD) as defined by DSM-IV criteria (except clause "does not occur exclusively during a mood disorder" of Criterion F for GAD) .
4. Subjects' bipolar symptoms must be no more than moderately severe, defined as a CGI-BP < 4.
5. Subjects' anxiety symptoms must be at least moderately severe, defined as a CGI-S > 4.
6. Subjects must not be receiving mood stabilizing, antidepressant, antipsychotic, or anxiolytic medication for > one week prior to baseline. Patients receiving fluoxetine or depot antipsychotics should be off these medications for > four weeks prior to baseline.
7. Subjects or their legally authorized representative must sign the Informed Consent Document after the nature of the trial has been fully explained.
8. If female, subjects must be:

   * postmenopausal,
   * surgically incapable of childbearing,
   * or practicing medically acceptable effective method(s) of contraception (e.g., hormonal methods, barrier methods, intrauterine device) for at least one month prior to study entry and throughout the study.

Exclusion Criteria:

1. Subjects who do not have lifetime bipolar disorder by DSM-IV-TR (text revision) criteria.
2. Subjects who do not have lifetime panic disorder or generalized anxiety disorder by DSM-IV-TR criteria.
3. Subjects who are receiving treatment with an antimanic or mood stabilizing medication (lithium, valproate, carbamazepine, or an antipsychotic), and in the investigators' judgment, require ongoing treatment with that medication.
4. Subjects whose bipolar symptoms are presently more than moderately severe (CGI-BP > 5).
5. Subjects whose anxiety symptoms are presently less than moderately severe (CGI < 3).
6. Subjects with clinically significant suicidal or homicidal ideation.
7. Subjects with current psychotic symptoms.
8. Subjects with a current DSM-IV Axis I diagnosis of delirium, dementia, amnesia, or other cognitive disorders; a DSM-IV diagnosis of a substance dependence disorder within the past six months; or a lifetime DSM-IV psychotic disorder (e.g., schizophrenia or schizoaffective disorder).
9. Subjects with serious general medical illnesses including hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, or hematologic disease as determined by the clinical judgment of the clinical investigator. Subjects with hypo- or hyperthyroidism unless stabilized on thyroid replacement > 3 months.
10. Subjects with a clinically significant abnormality in their prestudy physical exam, vital signs, EKG, or laboratory tests.
11. Subjects who are allergic to or who have demonstrated hypersensitivity to risperidone.
12. Women who are pregnant or nursing.
13. Subjects who have received an experimental drug or used an experimental device within 30 days.
14. Subjects who have a history of neuroleptic malignant syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2004-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Clinical Global Improvement-21 Anxiety scale (CGI-21 Anxiety) | weekly

SECONDARY OUTCOMES:
Hamilton Anxiety scale (HAM-A) | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. McElroy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Sheehan DV, McElroy SL, Harnett-Sheehan K, Keck PE Jr, Janavs J, Rogers J, Gonzalez R, Shivakumar G, Suppes T. Randomized, placebo-controlled trial of risperidone for acute treatment of bipolar anxiety. J Affect Disord. 2009 Jun;115(3):376-85. doi: 10.1016/j.jad.2008.10.005. Epub 2008 Nov 29. PMID 19042026